CLINICAL TRIAL: NCT00859898
Title: A Multicenter, Randomized, Double-Blind, Active Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin 10 mg in Combination With Metformin as Initial Therapy as Compared With Dapagliflozin 10 mg Monotherapy and Metformin Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: Study of Dapagliflozin in Combination With Metformin XR to Initiate the Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB102-034; Eudract #: 2008-007548-33
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Metformin; Dapagliflozin; Hypoglycemic Agents; Pharmacologic Actions; Physiological Effects of Drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dapagliflozin + Metformin XR (Experimental): Dapagliflozin: Tablets, Oral, 10 mg, once daily, 24 weeks
  Metformin XR: Tablets, Oral, up to 2000 mg, once daily, 24 weeks
  Interventions: Drug: Dapagliflozin; Drug: Metformin XR
- Dapagliflozin + Placebo (Experimental): Dapagliflozin: Tablets, Oral, 10 mg, once daily, 24 weeks.
  Placebo: Metformin HCl Modified Release matching placebo tablets, once daily, 24 weeks.
  Interventions: Drug: Dapagliflozin; Drug: metformin HCl Modified Release matching Placebo
- Metformin XR + Placebo (Active Comparator): Metformin XR: Tablets, Oral, 500 mg up to 2000 mg, once daily 24 weeks
  Placebo: Dapagliflozin matching placebo tablets once daily, 24 weeks
  Interventions: Drug: Metformin XR; Drug: dapagliflozin matching Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 10 mg, once daily, 24 weeks
  Other Names: Farxiga™
  Arms: Dapagliflozin + Metformin XR; Dapagliflozin + Placebo
Drug: Metformin XR — Tablets, Oral, up to 2000 mg, once daily, 24 weeks
  Other Names: Glucophage®
  Arms: Dapagliflozin + Metformin XR
Drug: Metformin XR — Tablets, Oral, 500 mg up to 2000 mg, once daily 24 weeks
  Other Names: Glucophage®
  Arms: Metformin XR + Placebo
Drug: dapagliflozin matching Placebo — Tablets
  Arms: Metformin XR + Placebo
Drug: metformin HCl Modified Release matching Placebo — Tablets
  Arms: Dapagliflozin + Placebo

SUMMARY:
The primary purpose of this study is to compare the change from baseline in hemoglobin A1C achieved with dapagliflozin 10 mg in combination with metformin XR as compared with metformin XR monotherapy and compared with Dapagliflozin monotherapy, after 24 weeks of oral administration of double-blind treatment. The safety of treatment with dapagliflozin will also be assessed in this study

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive males and females, >= 18 years old and

<= 77 years old, with type 2 diabetes mellitus

* Subjects must have central laboratory pre-randomization hemoglobin A1C >= 7.5 and <= 12.0%
* C-peptide >= 1.0 ng/mL (0.34 nmol/L)
* Body Mass Index <= 45 kg/m2
* Must be able to perform self monitoring of blood glucose

Exclusion Criteria:

* aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3X*upper limit of normal (ULN)
* Serum Total bilirubin >2 mg/dL (34.2 µmol/L)
* Creatinine kinase >3*ULN
* Serum creatinine >= 1.50 mg/dL (133 µmol/L) for male subjects, >= 1.40 mg/dL (124 µmol/L) for female subjects
* Calcium value outside of the central laboratory normal reference range
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncological, endocrine, psychiatric, or rheumatic diseases
* Urine albumin:creatinine ratio (UACR) >1800 mg/g (203.4 mg/mmol Cr)
* Severe uncontrolled hypertension defined as systolic blood pressure (SBP) >=180 mmHg and/or diastolic blood pressure (DBP) >=110 mmHg
* Hemoglobin >=11.0 g/dL (110 g/L) for men; hemoglobin >=10.0 g/dL (100 g/L) for women
* Positive for hepatitis B surface antigen
* Positive for anti-hepatitis C virus antibody
* History of diabetes insipidus
* History of diabetic ketoacidosis or hyperosmolar nonketotic coma
* Symptoms of poorly controlled diabetes that would preclude participation in this trial

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1093 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (107):
- United States (64):
  - International Institute Of Clinical Research, Ozark, Alabama
  - Clinical Research Advantage, Inc./Mesa Family Med Ctr, Pc, Tempe, Arizona
  - Clinical Research Advantage, Inc., Tempe, Arizona
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Encompass Clinical Research-North Coast, Encinitas, California
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Valley Research, Fresno, California
  - Del Rosario Medical Clinic, Inc., Huntington Park, California
  - Irvine Center For Clinical Research, Inc., Irvine, California
  - Pacific Sleep Medicine Services (Avastra Clinical Trials), Redlands, California
  - Orange County Research Center, Tustin, California
  - Lynn Institute Of The Rockies, Colorado Springs, Colorado
  - Radiant Research, Inc., Denver, Colorado
  - Clinical Therapeutics Corporation, Coral Gables, Florida
  - Nextphase Clinical Trials, Inc., Miami, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Lake Hartwell Family Medicine, Hartwell, Georgia
  - Middle Georgia Drug Study Center, Llc, Perry, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Provident Clinical Research, Addison, Illinois
  - Cedar Crosse Research Center, Chicago, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Physicians Research Group, Indianapolis, Indiana
  - Borgess Research Institute, Kalamazoo, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Clinilabs, Inc., New York, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - Community Health Care, Inc., Canal Fulton, Ohio
  - Holzer Clinic, Inc, Gallipolis, Ohio
  - Wells Institute For Health Awareness, Kettering, Ohio
  - Newark Physician Associates, Newark, Ohio
  - Daniel G. Williams, Md, Perrysburg, Ohio
  - Physician Research, Inc., Zanesville, Ohio
  - Gilbert Medical Research, Llc, Bethany, Oklahoma
  - Tulsa Clinical Research, Llc, Tulsa, Oklahoma
  - Integris Family Care Yukon, Yukon, Oklahoma
  - Williamette Valley Clinical Studies, Eugene, Oregon
  - Dingmans Medical, Dingmans Ferry, Pennsylvania
  - Integrated Medical Group Pc/Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Wellmon Family Practice, Shippensburg, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Southeastern Research Associates, Inc., Greenville, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Parkway Medical Group, Fayetteville, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Southwind Medical Specialists, Memphis, Tennessee
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - Endocrine Associates, Houston, Texas
  - Village Family Practice, Houston, Texas
  - Juno Research, Llc., Houston, Texas
  - Non-Invasive Cardiovascular, Pa, Houston, Texas
  - Excel Clinical Research, Houston, Texas
  - Texas Center For Drug Development, Houston, Texas
  - Midland Clinical Research Center, Midland, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - Covenant Clinical Research, Pa, San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - Avastra Clinical Trials, Midvale, Utah
  - Seven Corners Medical Center, Falls Church, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- India (9):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Aminjikarai, Chennai
  - Local Institution, Haryāna, Karnal
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Indore, Madhya Pradesh
  - Local Institution, Nagpur, Maharashtra
  - Local Institution, Chennai, Tamil Nadu
  - Local Institution, Ghaziabad, Uttar Pradesh
  - Local Institution, Jaipur
- Mexico (8):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Durango, Durango
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Morelia, Michioacan
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Veracruz, Veracruz
  - Local Institution, Mérida, Yucatán
- Puerto Rico (3):
  - Local Institution, Fajardo
  - Local Institution, Ponce
  - Local Institution, San Juan
- Russia (16):
  - Local Institution, Ekaterinaburg
  - Local Institution, Kemerovo
  - Local Institution, Krasnoyarsk
  - Local Institution, Moscov
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Novosibirsk
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Saratov
  - Local Institution, Smolensk
  - Local Institution, Tyumen
  - Local Institution, Vladimir
  - Local Institution, Volgograd
  - Local Institution, Voronezh
  - Local Institution, Yaroslavl
- South Korea (7):
  - Local Institution, Bucheon-si, Gyeonggi-do
  - Local Institution, Goyang-si, Gyeonggi-do
  - Local Institution, Guri-si, Gyeonggi-do
  - Local Institution, Sungnam, Gyeonggi-do
  - Local Institution, Daegu
  - Local Institution, Incheon
  - Local Institution, Seoul

REFERENCES:
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 13-April-2009 to 26-November-2009. Study completed 12-May-2010. Drug naive participants with Type 2 Diabetes Mellitus who had inadequate glycemic control with diet and exercise. Inadequate glycemic control was defined as a hemoglobin A1c (HbA1c) ≥ 7.5% and ≤ 12.0%.
Pre-assignment Details: Qualification: 660 completed: 28 administrative, 373 no longer met criteria, 1 lack of efficacy, 26 withdrew consent, 1 lost to follow up (LTF), 4 other. Lead-In: 649 entered; 641 completed/ randomized: 1 adverse event, 1 administrative, 4 no longer met criteria, 1 withdrew consent, 1 LTF. Treated 638: 1 LTF, 1 non-compliance, 1 withdrew consent.
Groups:
- Dapagliflozin: Dapagliflozin: Tablets, Oral, 10 mg, once daily, 24 weeks.
  Placebo: Metformin hydrochloride (HCl) Modified Release matching placebo tablets, once daily, 24 weeks.
- Metformin XR: Metformin XR: Tablets, Oral, 500 mg up to 2000 mg, once daily 24 weeks
  Placebo: Dapagliflozin matching placebo tablets once daily, 24 weeks
Period: Overall Study
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Started | 211 | 219 | 208
Completed | 183 | 188 | 181
Not Completed | 28 | 31 | 27
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Adverse Event | 4 | 9 | 8
Not completed — Withdrawal by Subject | 11 | 8 | 11
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 10 | 11 | 5
Not completed — poor/non-compliance | 2 | 0 | 0
Not completed — No longer meets criteria | 0 | 1 | 0
Not completed — non-specified | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who took at least one dose of double-blind study medication.
Groups:
- Dapagliflozin: Dapagliflozin: Tablets, Oral, 10 mg, once daily, 24 weeks
  Placebo: Metformin HCl Modified Release matching placebo tablets, once daily, 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR | Total
Number analyzed (Participants) | 211 | 219 | 208 | 638
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (10.13) | 51.1 (11.53) | 52.7 (10.38) | 51.6 (10.72)
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 190 | 192 | 181 | 563
  Greater than, equal to (>=) 65 and < 75 years | 21 | 24 | 25 | 70
  >= 75 years | 0 | 3 | 2 | 5
  Not Reported | 0 | 0 | 0 | 0
Age, Customized [Number; unit: participants] — Female age categorization less than equal to (<=) 50 years or greater than (>) 50 years.
  participants
    Female <= 50 years | 43 | 44 | 44 | 131
    Female > 50 years | 62 | 70 | 67 | 199
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 114 | 111 | 330
  Male | 106 | 105 | 97 | 308
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of participants
  Participants
    Hispanic or Latino | 34 | 34 | 35 | 103
    Not Hispanic or Latino | 54 | 63 | 54 | 171
    Unknown or Not Reported | 123 | 122 | 119 | 364
Race/Ethnicity, Customized [Number; unit: participants]
  White | 174 | 176 | 166 | 516
  Black/African American | 11 | 13 | 8 | 32
  Asian | 24 | 27 | 31 | 82
  Other Race | 2 | 3 | 3 | 8
Body Mass Index [Number; unit: participants] — Body Mass Index (BMI) was kilograms (kg) body weight divided by height in meters (m) squared (kg/m^2). Less than (<); Greater than, equal to (>=).
  participants
    < 25 kg/m^2 | 20 | 25 | 21 | 66
    >= 25 kg/m^2 - <27 kg/m^2 | 23 | 24 | 20 | 67
    >= 27 kg/m^2 - <30 kg/m^2 | 45 | 39 | 49 | 133
    >= 30 kg/m^2 | 123 | 131 | 118 | 372
Waist Circumference [Mean (Standard Deviation); unit: cm] — The participants waist was measured in centimeters (cm).
  cm | 104.33 (13.678) | 103.86 (12.805) | 103.03 (13.224) | 103.75 (13.225)
Hemoglobin A1c [Mean (Standard Deviation); unit: percent of hemoglobin] — Hemoglobin A1c (HbA1c) was reported as percent of hemoglobin.
  percent of hemoglobin | 9.09 (1.258) | 9.05 (1.279) | 9.05 (1.308) | 9.06 (1.280)
Total Body Weight [Mean (Standard Deviation); unit: kg] — Participants were weighed and weight recorded in kilograms (kg).
  kg | 88.43 (19.668) | 88.53 (19.334) | 87.24 (19.423) | 88.08 (19.452)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24 (Last Observation Carried Forward) - Randomized Treated Participants
Description: Adjusted mean change in HbA1c from baseline at Week 24 (or the last post-baseline measurement prior to Week 24 if no Week 24 assessment was available, ie, last observation carried forward (LOCF) was determined. HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the Qualification and Lead-In Periods and on Day 1 and Weeks 4, 8, 12, 16, 20, and 24 in the Double-Blind Period.
Time Frame: Week 24
Population: N= Number of randomized participants, who took at least 1 dose of double-blind study medication, with non-missing baseline and Week 24 (LOCF) values.
Measure: Mean (Standard Error); unit: Percent of hemoglobin
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 202 | 216 | 203
Percent of hemoglobin | -1.98 (0.0759) | -1.45 (0.0734) | -1.44 (0.0757)
Statistical Analysis 1: Comparison: Dapagliflozin + Metformin XR vs Dapagliflozin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Dapagliflozin 10 mg plus metformin XR treatment group had to be superior to both monotherapy treatment groups to be considered significant. Two-sided significance level at α=0.05; treatment group as an effect and the baseline HbA1c value as a covariate; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.74 to -0.32], Standard Error of Mean 0.1056
Statistical Analysis 2: Comparison: Dapagliflozin + Metformin XR vs Metformin XR; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; treatment group as an effect and the baseline HbA1c value as a covariate; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.75 to -0.33], Standard Error of Mean 0.1072
Statistical Analysis 3: Comparison: Dapagliflozin vs Metformin XR; Test type: Non-Inferiority or Equivalence — The non-inferiority of dapagliflozin 10 mg versus metformin XR was demonstrated when the upper limit of the two-sided 95% confidence interval of the difference in change in HbA1c from baseline to Week 24 (LOCF) between dapagliflozin 10 mg and metformin XR was less than 0.35%; ANCOVA; treatment group as an effect and the baseline value as a covariate; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.22 to 0.20], Standard Error of Mean 0.1054
Statistical Analysis 4: Comparison: Dapagliflozin vs Metformin XR; When testing for superiority, significance is claimed only if dapagliflozin 10 mg is superior to metformin XR; Test type: Superiority or Other; p = 0.9144, ANCOVA — two-sided significance level at α=0.05; treatment group as an effect and the baseline HbA1c value as a covariate; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.22 to 0.20], Standard Error of Mean 0.1054

2. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 (LOCF) - Randomized, Treated Participants
Description: Data after rescue medication was excluded from this analysis. FPG was measured as milligrams per deciliter (mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained during the Qualification and Lead-In Periods and on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 of the Double-Blind Period.
Time Frame: Week 24
Population: Number analyzed = Number of randomized participants, who took at least 1 dose of double-blind study medication, with non missing baseline and Week 24 (LOCF) values.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 209 | 216 | 207
mg/dL | -60.4 (2.533) | -46.4 (2.494) | -34.8 (2.545)
Statistical Analysis 1: Comparison: Dapagliflozin + Metformin XR vs Dapagliflozin; A hierarchical closed testing procedure was implemented to control the familywise type I error rate related to this endpoint at the two-sided 0.05 level. Statistical tests were only performed for a given secondary endpoint if all previous sequential tests versus that treatment group were also significant; Test type: Superiority or Other; p < 0.0001, ANCOVA — two-sided significance level at α=0.05. Dapagliflozin 10 mg plus metformin XR treatment group had to be superior to both monotherapy treatment groups to be considered significant; treatment group as an effect and the baseline value as a covariate; Mean Difference (Final Values) = -13.9, 95% CI 2-sided [-20.9 to -7.0], Standard Error of Mean 3.558
Statistical Analysis 2: Comparison: Dapagliflozin + Metformin XR vs Metformin XR; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; treatment group as an effect and the baseline value as a covariate; Mean Difference (Final Values) = -25.5, 95% CI 2-sided [-32.6 to -18.5], Standard Error of Mean 3.590
Statistical Analysis 3: Comparison: Dapagliflozin vs Metformin XR; Test type: Non-Inferiority or Equivalence — The non-inferiority of dapagliflozin 10 mg versus metformin XR was demonstrated when the upper limit of the two-sided 95% confidence interval of the difference in change FPG from baseline to Week 24 (LOCF) between dapagliflozin 10 mg and metformin XR was less than 15 mg/dL; ANCOVA; treatment group as an effect and the baseline value as a covariate; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-18.6 to -4.6], Standard Error of Mean 3.566
Statistical Analysis 4: Comparison: Dapagliflozin vs Metformin XR; When testing for superiority, significance is claimed only if dapagliflozin 10 mg is superior to metformin XR; Test type: Superiority or Other; p = 0.0012, ANCOVA — two-sided significance level at α=0.05; treatment group as an effect and the baseline value as a covariate; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-18.6 to -4.6], Standard Error of Mean 3.566

3. Secondary Outcome: Percent Adjusted for Baseline HbA1c of Participants Achieving a Therapeutic Glycemic Response at Week 24 (LOCF) - Randomized, Treated Participants
Description: Therapeutic glycemic response was defined as HbA1c less than 7.0%. n=Number of participants with HBA1c less than (<) 7 % at Week 24, last observation carried forward (LOCF) while N=number of randomized participants with non-missing baseline and Week 24 (LOCF) values. Percent=n/N and was adjusted for Baseline HbA1c. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin.
Time Frame: Week 24
Population: N=number of randomized participants with non-missing baseline and Week 24 (LOCF) values; N=202, 216, 203, respectively. n=number of responders: 92, 69, 72, respectively. n/N=percent. Percent is then adjusted for baseline HbA1c.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 202 | 216 | 203
Percent of participants | 46.6 [40.1 to 53.0] | 31.7 [25.7 to 37.7] | 35.5 [28.8 to 41.7]
Statistical Analysis 1: Comparison: Dapagliflozin + Metformin XR vs Dapagliflozin; The probability of response was modeled using a logistic regression model with baseline HbA1c as the covariate. Treatment group estimates of response rate were then obtained by integrating each group's modeled probability of response over the observed distribution of baseline covariate (combined across groups); Test type: Superiority or Other; p = 0.0012, Regression, Logistic — Dapagliflozin 10 mg plus metformin XR treatment group had to be superior to both monotherapy treatment groups to be considered significant; Logistic regression based on the methodology of Zhang, Tsiatis and Davidian and Tsiatis, Davidian, Zhang and Lu, with adjustment for baseline HbA1c; Mean Difference (Final Values) = 14.9, 95% CI 2-sided [5.9 to 23.9], Standard Error of Mean 4.598
Statistical Analysis 2: Comparison: Dapagliflozin + Metformin XR vs Metformin XR; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0165, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 11.3, 95% CI 2-sided [2.1 to 20.6], Standard Error of Mean 4.730

4. Secondary Outcome: Adjusted Mean Change From Baseline in HbA1C at Week 24 (LOCF) in Participants Whose Baseline HbA1C Category ≥9.0%
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. The population included those randomized, treated participants whose Baseline HbA1c was greater than, equal to (>=) 9.0%. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: Week 24
Population: N= Number of randomized participants, who took at least 1 dose of double-blind study medication, with non missing baseline and Week 24 (LOCF) values, whose baseline HbA1c was >=9.0%.
Measure: Mean (Standard Error); unit: Percent of Hemoglobin
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 106 | 97 | 95
Percent of Hemoglobin | -2.59 (0.1249) | -2.14 (0.1305) | -2.05 (0.1318)
Statistical Analysis 1: Comparison: Dapagliflozin + Metformin XR vs Dapagliflozin; A hierarchical closed testing procedure was implemented to control the familywise type I error rate related to this endpoint at the two-sided 0.05 level. Statistical testing was only performed if the dapagliflozin 10 mg plus metformin XR group was statistically significantly superior to both control groups for the primary efficacy endpoint. Tests were only performed for a given secondary endpoint if all previous sequential tests versus that treatment group were also significant; Test type: Superiority or Other; p = 0.0133, ANCOVA — [p-value comment as in outcome 2, analysis 1]; : treatment group as an effect and the baseline HbA1c value as a covariate; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.81 to -0.09], Standard Error of Mean 0.1807
Statistical Analysis 2: Comparison: Dapagliflozin + Metformin XR vs Metformin XR; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0036, ANCOVA — [p-value comment as in outcome 2, analysis 1]; treatment group as an effect and the baseline HbA1c value as a covariate; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.89 to -0.18], Standard Error of Mean 0.1817

5. Secondary Outcome: The Adjusted Mean Change From Baseline in Total Body Weight at Week 24 (LOCF) - Randomized, Treated Participants
Description: Adjusted mean change from baseline in total body weight at Week 24 (or the last post-baseline measurement prior to Week 24 if no Week 24 assessment was available was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight was measured in kilograms (kg). Body weight measurements were obtained during the Qualification and Lead-In Periods and on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 of the Double-Blind Period.
Time Frame: Week 24
Population: N= Number of randomized participants, who took at least 1 dose of double-blind study medication, with non missing baseline and Week 24 (LOCF) values.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 209 | 219 | 208
kg | -3.33 (0.2401) | -2.73 (0.2346) | -1.36 (0.2408)
Statistical Analysis 1: Comparison: Dapagliflozin + Metformin XR vs Metformin XR; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — two-sided significance level at α=0.05; treatment group as an effect and the baseline value as a covariate; Mean Difference (Final Values) = -1.97, 95% CI 2-sided [-2.64 to -1.30], Standard Error of Mean 0.3401
Statistical Analysis 2: Comparison: Dapagliflozin vs Metformin XR; Statistical tests were only performed for a given secondary endpoint if all previous sequential tests versus that treatment group were also significant; Test type: Superiority or Other; p < 0.0001, ANCOVA — two-sided significance level at α=0.05; treatment group as an effect and the baseline value as a covariate; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-2.03 to -0.71], Standard Error of Mean 0.3362

6. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Discontinuation Due to AEs, During the 12 Week Double Blind Period, Including Data After Rescue - All Treated Participants
Description: Medical Dictionary for Regulatory Activities (MedDRA), version 12.1 AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug as per the investigator. Events captured from baseline to last dose plus 4 days for AEs, plus 30 days for SAEs during the Double Blind 12 Week Period. Data after rescue included.
Time Frame: Day 1 of Double Blind Period to end of Week 24 Plus 30 days
Population: Participants who received at least 1 dose of double-blind study medication during the double-blind treatment period. Data after rescue were also included.
Measure: Number; unit: participants
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 211 | 219 | 208
participants
  Adverse Event (AE) | 126 | 132 | 118
  Related Adverse Event | 34 | 47 | 32
  Serious Adverse Event (SAE) | 3 | 5 | 4
  Related SAE | 0 | 1 | 1
  Discontinued due to AE | 4 | 9 | 8
  Deaths | 0 | 0 | 1
  Discontinued due to SAE | 0 | 1 | 1

7. Secondary Outcome: Number of Participants With Adverse Events of Special Interest During the 12 Week Double Blind Period - All Treated Participants
Description: Participants with AEs of hypoglycemia, cardiac/vascular disorders, renal impairment or failure, volume depletion (hypotension/dehydration/hypovolemia), fractures, urinary stones, and other reports suggestive of genital infection or urinary tract infection (UTI) were summarized using MedDRA version 13.0. Data after rescue included for all special AEs except hypoglycemia (excluded data after rescue). Major hypoglycemic episode: symptomatic requiring 3rd party assistance due to severe impairment in consciousness or behavior with a glucose value < 54 mg/dL and prompt recovery after glucose/glucagon; Minor: either symptomatic with glucose measurement < 63 mg/dL, regardless of need for 3rd party assistance, or asymptomatic with glucose < 63 mg/dL that does not qualify as major; Other: suggestive but not meeting criteria for major or minor.
Time Frame: Baseline to last dose plus 4 days in 12 Week Double Blind Period
Population: Randomized participants who received at least one dose of study medication in the double-blind period. Data after rescue included for all AEs except hypoglycemia, which excluded data after rescue.
Measure: Number; unit: participants
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 211 | 219 | 208
participants
  Cardiac Disorder AEs | 3 | 3 | 5
  Vascular Disorder AEs | 4 | 10 | 8
  Hypoglycemia AEs (excluding data after rescue) | 7 | 2 | 6
  Hypoglycemia Major Episode | 0 | 0 | 0
  Hypoglycemia Minor Episode | 1 | 0 | 1
  Hypoglycemia Other Episode | 6 | 2 | 5
  AEs Suggestive of Genital Infection | 18 | 28 | 5
  AEs Suggestive of UTI | 16 | 24 | 9
  AEs of Renal Impairment or Failure | 2 | 4 | 1
  AEs of Hypotension | 0 | 1 | 0
  AEs of Syncope | 0 | 1 | 0
  AEs of Fracture | 2 | 1 | 0
  AEs of Urinary Stones | 0 | 0 | 1

8. Secondary Outcome: Mean Change From Baseline in Seated Systolic and Diastolic Blood Pressure at Week 24 - Treated Participants
Description: Measurements were taken during the Qualification and Lead-In Periods and on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 in the Double Blind Period. Blood pressure values were obtained: after the participant was seated quietly for 5 minutes; at least 8 hours after the last ingestion of caffeine, alcohol, or nicotine; and in the same arm (right or left) consistently through out the study. Systolic and Diastolic pressures were measured in millimeters of mercury (mmHg). Data after rescue were also included. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: Week 24
Population: N=number of participants who took at least 1 dose of double-blind study medication, with non missing baseline and Week 24 values.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 182 | 185 | 179
mmHg
  Systolic (N=182, 185, 179) | -3.3 (0.947) | -4.0 (0.883) | -1.2 (1.010)
  Diastolic (N=182, 185, 179) | -1.8 (0.579) | -1.9 (0.525) | 0.0 (0.606)

9. Secondary Outcome: Mean Change From Baseline in Seated Heart Rate at Week 24 - Randomized, Treated Participants
Description: Measurements were taken during the Qualification and Lead-In Periods and on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 in the Double Blind Period. Heart rate values were obtained: after the participant was seated quietly for 5 minutes; at least 8 hours after the last ingestion of caffeine, alcohol, or nicotine; and in the same arm (right or left) consistently throughout the study. Heart rate was measured in beats per minute (bpm). Data after rescue were also included. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: Week 24
Population: as for outcome 8
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 182 | 185 | 179
bpm | 0.6 (0.607) | -0.1 (0.593) | 0.5 (0.594)

10. Secondary Outcome: Number of Participants With Normal or Abnormal Electrocardiogram Summary Tracing at Week 24 (LOCF) - Randomized, Treated Participants
Description: 12-Lead electrocardiograms (ECGs) were performed at entry into Lead-In Period Day -7 visit and Week 24/End of treatment visit (last observation carried forward) on participants who were supine. ECGs were assessed by the investigator. Baseline (BL) was Day -7 for this parameter. Data after rescue included.
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 211 | 219 | 208
participants
  Normal at BL, Normal at Week 24 (N=211, 219, 208) | 101 | 107 | 94
  Abnormal BL, Normal at Week 24 (N=211, 219, 208) | 15 | 13 | 22
  Normal BL, Abnormal at Week 24 (N=211, 219, 208) | 18 | 8 | 9
  Abnormal BL, Abnormal at Week 24 (N=211, 219, 208) | 53 | 68 | 59
  Normal at BL, Not Reported at Week 24 | 19 | 15 | 15
  Abnormal at BL, Not Reported at Week 24 | 5 | 8 | 8
  Not Reported at BL, Abnormal at Week 24 | 0 | 0 | 1

11. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities (Not Including Liver Function) in 24 Week Double Blind Treatment Period, Including Data After Rescue - Randomized, Treated Participants
Description: Laboratory samples: Qualification and Lead-In Periods, Day 1, Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 of Double-Blind Period. Baseline (BL)=last assessment prior to start of first dose of double-blind study medication. Data after rescue included. Pretreatment (PreRX); grams per deciliter (g/dL); upper limit of normal (ULN); milliequivalent per liter (mEq/L); Units per liter (U/L), blood urea nitrogen (BUN). Marked abnormality Low (High) defined: hemoglobin <6 (>18 females or >20 males) g/dL; hematocrit <20% ( >55% females or >60% males); creatinine (>=1.5*preRX, >=2.5 mg/dL); glucose <54 (>350) mg/dL; creatine kinase (>5*ULN);calcium <7.5 (>=1 mg/dL from ULN and >= 0.5mg/dL from PreRX); sodium <130 or < 120 male/female (>150 mEq/L; potassium <=2.5 (>=6.0) mEq/L; bicarbonate <= 13 mEq/L; inorganic phosphorus: <=1.8 if age 17-65 or <=2.1 if age >=66, (>=5.6 if age 17-65 or >=5.1) mg/dL if age >=66; albumin <=2 (>6) g/dL; urine albumin(alb) / creatinine (creat) ratio (>1800 mg/g)
Time Frame: Baseline to Week 24/end of treatment plus 4 days
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 209 | 218 | 207
participants
  Hematocrit High > 55% (N=209, 218, 206) | 1 | 4 | 1
  Hemoglobin High >18 g/dL(N=209, 218, 207) | 5 | 4 | 1
  Creatinine >1.5*PreRX (N=209, 218, 207) | 8 | 2 | 5
  Glucose High > 350 mg/dL (N=209, 218, 207) | 1 | 2 | 3
  Albumin low or high (N=209, 218, 207) | 0 | 0 | 0
  Calcium Low <7.5mg/dL (N=209, 218, 207) | 1 | 2 | 1
  Calcium High >=1mg/dL+ULN (N=209, 218, 207) | 0 | 2 | 0
  Bicarbonate Low <=13mEq/L (N=209, 218, 207) | 3 | 0 | 0
  Potassium High >=6 mEq/L (N=209, 218, 207) | 2 | 3 | 6
  Sodium Low <130 mEq/L (N=209, 218, 207) | 2 | 2 | 2
  Sodium High >150 mEq/L (N=209, 218, 207) | 5 | 5 | 2
  Sodium Low <120 mEq/L (N=209, 218, 207) | 0 | 1 | 0
  inorganic phosphorus (high)(N=209, 218, 207) | 7 | 13 | 3
  Urine albumin/creat ratio (high)(N=209, 218, 206) | 0 | 3 | 1

12. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Liver Function in 24 Week Double Blind Treatment Period, Including Data After Rescue - Randomized, Treated Participants
Description: Safety laboratory measurements were obtained during the Qualification and Lead-In Periods and on Day 1 of the Double-Blind Period and at Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24. BL was defined as the last assessment prior to the start of the first dose of the double-blind study medication. Data included from BL up to and including the last day of treatment plus 30 days. Liver function abnormality criteria: FDA Guidance for Industry: Premarketing Clinical Evaluation (July 2009). Data after rescue was also included. Abbreviations: Pretreatment (PreRX), upper limit of normal (ULN); greater than (>) less than (<); Units per liter (U/L), alanine aminotransferase (ALT); aspartate aminotransferase (AST); alkaline phosphatase (ALP). Marked abnormality Low (High) defined: ALP, AST and ALT (>3*ULN); bilirubin (>2*ULN if PreRX <= ULN; >3*ULN if PreRX > ULN); AST or ALT plus (+) bilirubin elevation: AST or ALT >3*ULN and bilirubin >1.5*ULN within 14 days on or after ALT elevation.
Time Frame: Baseline to Week 24/end of treatment plus 30 days
Measure: Number; unit: participants
Arm/Group | Dapagliflozin + Metformin XR | Dapagliflozin | Metformin XR
Number analyzed (Participants) | 210 | 219 | 208
participants
  AST >3*ULN (N=210, 219, 208) | 2 | 3 | 2
  AST >5*ULN (N=210, 219, 208) | 0 | 1 | 1
  ALT >3*ULN (N=210, 219, 208) | 2 | 4 | 7
  ALT >5*ULN (N=210, 219, 208) | 0 | 1 | 2
  ALT >10*ULN (N=210, 219, 208) | 0 | 0 | 1
  AST or ALT > 3*ULN (N=210, 219, 208) | 3 | 5 | 7
  AST or ALT > 5*ULN (N=210, 219, 208) | 0 | 1 | 2
  AST or ALT > 10*ULN (N=210, 219, 208) | 0 | 0 | 1
  Total bilirubin >1.5*ULN (N=210, 219, 207) | 0 | 2 | 1
  AST or ALT + Bilirubin (High) (N=210, 219, 208) | 0 | 0 | 1
  ALP >1.5*ULN (N=210, 219, 208) | 5 | 4 | 3
  ALP >3*ULN (N=210, 219, 208) | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 24 Weeks plus 30 days; Day 1 of double blind treatment to last patient, last visit.
Arm/Group | Dapagliflozin | Dapagliflozin + Metformin XR | Metformin XR
Serious Adverse Events (participants affected / at risk) | 5/219 | 3/211 | 4/208
Other Adverse Events (participants affected / at risk) | 32/219 | 26/211 | 24/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin (N=219) | Dapagliflozin + Metformin XR (N=211) | Metformin XR (N=208)
Lung abscess (Infections and infestations) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 2
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin (N=219) | Dapagliflozin + Metformin XR (N=211) | Metformin XR (N=208)
Diarrhoea (Gastrointestinal disorders) | 6 | 15 | 20
Urinary tract infection (Infections and infestations) | 17 | 6 | 4
Vulvovaginal mycotic infection (Infections and infestations) | 11 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.